CLINICAL TRIAL: NCT00753675
Title: A Randomized, Multicentre, Phase II, Parallel-Group Trial of Vandetanib Monotherapy or Vandetanib in Combination With Gemcitabine Versus Gemcitabine Plus Vandetanib Matching Placebo in Subjects With Advanced Biliary Tract Cancer (Gallbladder Cancer, Cancer of the Extrahepatic Bile Duct, Intrahepatic Cholangiocarcinoma and Ampullary Carcinoma)
Brief Title: Vandetanib Gemcitabine Or Placebo Plus Gemcitabine Or Vandetanib Monotherapy In Advanced Biliary Tract Cancer
Acronym: VANGOGH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4200L00007; EUDRACT n° 2007-003056-12
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Biliary Tract Cancer; Gallbladder Cancer; Cancer Of The Extrahepatic Bile Duct; Ampullary Carcinoma
Keywords: Intrahepatic; Cholangiocarcinoma; Vandetanib; Zactima; Advanced; Biliary; Tract; Gallbladder; Extrahepatic Bile Duct; Intrahepatic Cholangiocarcinoma; Ampullary Carcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms; Cholangiocarcinoma | interventions — vandetanib; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Vandetanib 300 mg as a once daily oral dose, from Day 1
  Interventions: Drug: ZD6474, Vandetanib
- B (Experimental): Gemcitabine administered intravenously at 1000 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg orally once-daily, from Day 1 (after 6 cycles, in the absence of disease progression or unacceptable toxicity, Investigators remain at liberty to continue Gemcitabine plus Vandetanib / Placebo or to continue Vandetanib / Placebo monotherapy)
  Interventions: Drug: ZD6474, Vandetanib; Drug: Gemcitabine
- C (Placebo Comparator): Gemcitabine administered intravenously at 1000 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to 6 cycles plus Vandetanib 100 mg Matching Placebo orally once-daily, from Day 1 (after 6 cycles, in the absence of disease progression or unacceptable toxicity, Investigators remain at liberty to continue Gemcitabine plus Vandetanib / Placebo or to continue Vandetanib / Placebo monotherapy).
  Interventions: Drug: Gemcitabine; Drug: Placebo matching ZD6474

INTERVENTIONS:
Drug: ZD6474, Vandetanib — 300 mg as a once daily oral dose, from Day 1 until disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Other Names: Zactima
  Arms: A
Drug: ZD6474, Vandetanib — 100 mg as a once daily oral dose, from Day 1 until disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Other Names: Zactima
  Arms: B
Drug: Gemcitabine — administered intravenously at 1000 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to 6 cycles or until disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Other Names: Gemzar
  Arms: B; C
Drug: Placebo matching ZD6474 — Placebo to match ZD6474 100 mg as a once daily oral dose, from Day 1 until disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Arms: C

SUMMARY:
The primary objective of the trial is to determine the efficacy of VANDETANIB monotherapy or VANDETANIB plus GEMCITABINE or PLACEBO plus GEMCITABINE in prolonging the progression-free survival (PFS) at the trial closure in patients with advanced (unresectable or metastatic) biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed advanced (unresectable or metastatic) biliary tract cancer (gallbladder cancer, cancer of the extrahepatic bile duct, intrahepatic cholangiocarcinoma and ampullary carcinoma)
* Patients must have measurable or evaluable but non-measurable disease
* Chemotherapy-naïve (prior chemotherapy in the adjuvant setting completed more than 3 months before the trial entry is accepted).
* WHO performance status 0 to 2: patients must have a WHO PS ≤ 2

Exclusion Criteria:

* Patients must not have received prior systemic therapy for advanced (unresectable or metastatic) disease; prior chemotherapy in the adjuvant setting within 3 months before the trial entry is accepted
* Inadequate end-organ function or Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance wit
* Significant cardiovascular event (e.g. myocardial infarction, superior vena cava [SVC] syndrome, New York Heart Association [NYHA] classification of heart disease ³2) within 3 months before entry, or presence of cardiac disease that in the opinion of
* History of arrhythmia or QTc with Bazett's correction unmeasurable or ≥ 480 msec on screening ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2008-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Italy (15):
  - Research Site, Brescia, BS
  - Research Site, Florence, FI
  - Research Site, Genova, GE
  - Research Site, Milan, Mi
  - Research Site, Palermo, PA
  - Research Site, Aviano, PN
  - Research Site, Parma, PR
  - Research Site, Reggio Emilia, RE
  - Research Site, Ancona
  - Research Site, Livorno
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Ravenna
  - Research Site, Rho
  - Research Site, Torino

REFERENCES:
- [Background] Wedge SR, Ogilvie DJ, Dukes M, Kendrew J, Chester R, Jackson JA, Boffey SJ, Valentine PJ, Curwen JO, Musgrove HL, Graham GA, Hughes GD, Thomas AP, Stokes ES, Curry B, Richmond GH, Wadsworth PF, Bigley AL, Hennequin LF. ZD6474 inhibits vascular endothelial growth factor signaling, angiogenesis, and tumor growth following oral administration. Cancer Res. 2002 Aug 15;62(16):4645-55. PMID 12183421
- [Derived] Santoro A, Gebbia V, Pressiani T, Testa A, Personeni N, Arrivas Bajardi E, Foa P, Buonadonna A, Bencardino K, Barone C, Ferrari D, Zaniboni A, Tronconi MC, Carteni G, Milella M, Comandone A, Ferrari S, Rimassa L. A randomized, multicenter, phase II study of vandetanib monotherapy versus vandetanib in combination with gemcitabine versus gemcitabine plus placebo in subjects with advanced biliary tract cancer: the VanGogh study. Ann Oncol. 2015 Mar;26(3):542-7. doi: 10.1093/annonc/mdu576. Epub 2014 Dec 23. PMID 25538178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 180 subjects were screened at 19 sites and 174 were randomized
Groups:
- Arm A Vandetanib 300 mg: Vandetanib 300 mg as a once daily oral dose, from Day 1
- Arm B Vandetanib 100mg + Gemcitab: Gemcitabine administered intravenously at 1000 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to plus Vandetanib 100 mg orally once-daily, from Day 1 (after 6 cycles, in the absence of disease progression or unacceptable toxicity, Investigators remain at liberty to continue Gemcitabine plus Vandetanib / Placebo or to continue Vandetanib / Placebo monotherapy)
- ARM C Placebo+ Gemcitabine: Gemcitabine administered intravenously at 1000 mg/m2 over 30 minutes on Days 1 and 8 of each 21-day cycle up to 6 cycles plus Vandetanib 100 mg Matching Placebo orally once-daily, from Day 1 (after 6 cycles, in the absence of disease progression or unacceptable toxicity, Investigators remain at liberty to continue Gemcitabine plus Vandetanib / Placebo or to continue Vandetanib / Placebo monotherapy).
Period: Overall Study
Arm/Group | Arm A Vandetanib 300 mg | Arm B Vandetanib 100mg + Gemcitab | ARM C Placebo+ Gemcitabine
Started | 59 | 59 | 56
Completed | 0 | 0 | 0
Not Completed | 59 | 59 | 56
Not completed — other reason | 11 | 12 | 13
Not completed — Death | 1 | 2 | 4
Not completed — Adverse Event | 11 | 9 | 4
Not completed — Objective progression of disease | 35 | 35 | 35
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patient screened 180 Patient Randomized 174 (1 never treated) Sceening failures 6 Patient Treated 173 (ITT=165 ; 8 excluded from ITT due to missing postbaseline assesment)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Vandetanib 300 mg | Arm B Vandetanib 100mg + Gemcitab | ARM C Placebo+ Gemcitabine | Total
Number analyzed (Participants) | 59 | 58 | 56 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Population
  years | 62.39 (10.108) | 64.41 (9.455) | 63.95 (8.764) | 63.57 (9.456)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population
  Participants
    Female | 34 | 27 | 31 | 92
    Male | 25 | 31 | 25 | 81

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression was defined as Time from the date of first dose of study medication to progression of disease, or death (it also includes patients who are lost to follow-up or have withdrawn consent) and evaluated with RECIST criteria as an increase of at least 20% in the sum of longest diameter (LD) of target lesion(s) taking as reference the smallest sum of LD since the treatment started or any new lesion(s).
Time Frame: up to 1032 days
Population: ITT
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A Vandetanib 300 mg | Arm B Vandetanib 100mg + Gemcitab | ARM C Placebo+ Gemcitabine
Number analyzed (Participants) | 56 | 57 | 52
days | 105 [72 to 155] | 114 [91 to 193] | 148 [72 to 225]

2. Secondary Outcome: Objective Tumor Response Rate (CR+PR),
Description: Objective Tumor Response Rate was defined as complete response (CR) + partial response (PR) evaluated by RECIST. CR was defined as disappearance of all target lesions. PR was defined as at least 30% decrease in the sum of longest diameters (LD) of target lesion(s) taking as reference the baseline sum of LD
Time Frame: up to 1032 days
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Arm A Vandetanib 300 mg | Arm B Vandetanib 100mg + Gemcitab | ARM C Placebo+ Gemcitabine
Number analyzed (Participants) | 56 | 57 | 52
Participants
  Objective Response = NO | 54 | 46 | 45
  Objective Response = YES | 2 | 11 | 7

3. Secondary Outcome: Disease Control Rate (CR+PR+SD)
Description: DCR is the sum of patients with a best overall CR, PR or SD (>=8 weeks) by the patient in the analysis
Time Frame: up to 1032 days
Population: ITT
Measure: Number; unit: Partecipants
Arm/Group | Arm A Vandetanib 300 mg | Arm B Vandetanib 100mg + Gemcitab | ARM C Placebo+ Gemcitabine
Number analyzed (Participants) | 56 | 57 | 52
Partecipants
  Disease control rate = NO | 42 | 40 | 32
  Disease control rate = YES | 14 | 17 | 20

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined from the date of first documentation of response until date of PD or death
Time Frame: up to 1032 days
Population: ITT (best response of CR or PR only)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A Vandetanib 300 mg | Arm B Vandetanib 100mg + Gemcitab | ARM C Placebo+ Gemcitabine
Number analyzed (Participants) | 2 | 11 | 7
Days | 277 [267 to 286] | 179 [85 to 369] | 127 [85 to 152]

5. Secondary Outcome: Overall Survival
Description: OS is defined from the date of randomization to death
Time Frame: up to 1032 days
Population: ITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A Vandetanib 300 mg | Arm B Vandetanib 100mg + Gemcitab | ARM C Placebo+ Gemcitabine
Number analyzed (Participants) | 56 | 57 | 52
Days | 228 [190 to 364] | 284 [213 to 359] | 307 [254 to 523]

ADVERSE EVENTS:
Arm/Group | Arm A Vandetanib 300 mg | Arm B Vandetanib 100mg + Gemcitab | ARM C Placebo+ Gemcitabine
Serious Adverse Events (participants affected / at risk) | 16/59 | 15/58 | 12/56
Other Adverse Events (participants affected / at risk) | 57/59 | 53/58 | 50/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A Vandetanib 300 mg (N=59) | Arm B Vandetanib 100mg + Gemcitab (N=58) | ARM C Placebo+ Gemcitabine (N=56)
Disseminated Intravascular (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood Bilirubin (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2) | 0/0 (0) | 0/0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Torsade de Pointes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Duodenal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Condition Aggravated (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 2 (2)
Cholangites (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubineamia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2)
Blood Bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Repolarisation Abnormaly (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Vandetanib 300 mg (N=59) | Arm B Vandetanib 100mg + Gemcitab (N=58) | ARM C Placebo+ Gemcitabine (N=56)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 10 (20) | 7 (18)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Asthenia (General disorders) | 7 (7) | 14 (17) | 15 (20) — General disorders and administration site conditions
Acute Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (5)
Agitated Depression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep Vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dessemintaed Intracascula Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubineamia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Iron deficency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukcytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 6 (17)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet production decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 5 (7) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (15) | 10 (28)
Arrhytmia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (2) | 1 (1)
Bundle branch block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle Branch block right (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diabete Mellitus (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycamia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular icterus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Periorbital Oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 15 (16) | 8 (9) | 14 (17)
Abdominal Pain upper (Gastrointestinal disorders) | 3 (3) | 6 (6) | 6 (6)
Aborectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 15 (32) | 6 (13) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4)
Dyshagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 6 (7) | 17 (29)
Oral Mucosal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pelvic Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 8 (11) | 5 (7) | 9 (21)
Chest Pain (General disorders) | 3 (3) | 2 (2) | 1 (2)
Chills (General disorders) | 1 (1) | 1 (2) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 8 (9) | 7 (9) | 8 (11)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gravitational oedema (General disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperhidrosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 4 (4) | 4 (6) | 0 (0)
Multi organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 3 (3)
Oedema Peripheral (General disorders) | 2 (2) | 3 (9) | 1 (3)
Pain (General disorders) | 2 (2) | 3 (4) | 1 (2)
Pyrexia (General disorders) | 8 (10) | 14 (22) | 14 (22)
Ascites (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangites (Hepatobiliary disorders) | 3 (3) | 2 (3) | 3 (3)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (10) | 5 (10) | 3 (3)
Hypertrasaminasaemia (Hepatobiliary disorders) | 2 (3) | 2 (2) | 2 (2)
Hypoalbuminaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (3) | 3 (3) | 3 (3)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Cystis escherichia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth abcess (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Aspartate aminotranferase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Asparteate amonotranferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood Bilirubin (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Bilirubin increased (Investigations) | 3 (5) | 1 (1) | 0 (0)
Blood creatine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehdrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 2 (2) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 2 (3) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormaly (Investigations) | 1 (1) | 1 (1) | 0 (0)
Gamma -glumayltransferase (Investigations) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (2) | 3 (5)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminase increased (Investigations) | 1 (2) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 8 (10) | 4 (4)
Deydratation (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in the extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal Compression Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Clonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Head Discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5)
Hypogeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 2 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder due to general medical condition , insomnia type (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (5) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercreatininaemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (5)
Renal failure (Renal and urinary disorders) | 2 (2) | 3 (4) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Strangury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysponea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 4 (4)
Dysponea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Metastic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (8) | 3 (4) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 5 (13) | 4 (4) | 4 (5)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Face Oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 15 (21) | 5 (5) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Toxicity (Skin and subcutaneous tissue disorders) | 2 (6) | 3 (3) | 1 (1)
Diastolic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 14 (17) | 9 (10) | 4 (6)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Urine colour abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.